CLINICAL TRIAL: NCT07317596
Title: Efficacy of Methylprednisolone and Hyaluronic Acid, Individually and in Combination, on Reducing Postoperative Complications After Mandibular Third Molar Extraction
Brief Title: Comparing Methylprednisolone And Hyaluronic Acid To Reduce Wisdom Tooth Surgery Complications
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Amal Yahya Mohammed Al-Eryani, Maxillofacial Surgeon, Sana'a University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 742
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Wisdom Tooth Removal; Post Operative Complications; Hyaluronic Acid; Methylprednisolone
Keywords: Mandibular third molar; Surgical extraction; Complications; Efficacy; Hyaluronic acid; Methylprednisolone
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (No Intervention): The control group will receive neither hyaluronic acid nor methylprednisolone
- Hyaluronic acid only (Experimental): Hyaluronic acid placement only
  Interventions: Biological: Hyaluronic Acid (HA)
- Methylprednisolone only (Experimental): Methylprednisolone injection only
  Interventions: Drug: Methyl Prednisolone (MP)
- Combination (Experimental): Methylprednisolone + Hyaluronic acid
  Interventions: Drug: Methyl Prednisolone (MP); Biological: Hyaluronic Acid (HA)

INTERVENTIONS:
Drug: Methyl Prednisolone (MP) — Methylprednisolone sodium succinate is a synthetic glucocorticoid (corticosteroid) administered intravenously at a single dose of 125 mg one hour prior to the surgical extraction of the impacted mandibular third molar. The purpose of this intervention is to reduce the inflammatory response, thereby controlling post-operative complications such as pain, swelling (edema), and limited mouth opening (trismus).
  Arms: Combination; Methylprednisolone only
Biological: Hyaluronic Acid (HA) — Hyaluronic acid (HA) is a naturally occurring glycosaminoglycan that is placed directly into the tooth socket after the surgical extraction of the impacted mandibular third molar. A volume of 2 ml of HA is applied before the surgical site is closed. This intervention is intended to promote tissue healing, reduce inflammation, and aid in the control of post-operative pain and swelling.
  Arms: Combination; Hyaluronic acid only

SUMMARY:
The goal of this clinical trial is to assess and compare the effectiveness of methylprednisolone and hyaluronic acid (HA), alone and in combination, in managing post-operative complications following the surgical extraction of impacted mandibular third molars (wisdom teeth). It will also learn about the safety and side effects of these treatments.

The main questions it aims to answer are:

* How effectively does methylprednisolone reduce post-operative pain, swelling (edema), and limited mouth opening (trismus)?
* How effectively does hyaluronic acid reduce post-operative pain, swelling (edema), and limited mouth opening (trismus)?
* Is the combination of methylprednisolone and hyaluronic acid more effective than either treatment alone in controlling these post-operative complications?
* What complications (e.g., soft tissue issues, infection) do participants experience with each treatment group? Researchers will compare the effects of methylprednisolone (given intravenously before surgery), hyaluronic acid (placed in the tooth socket after extraction), and a combination of both, against a control group that receives standard care (saline irrigation) to see which treatment or combination is most effective.

Participants will be medically healthy adults between the ages of 18 and 40 who are undergoing the surgical extraction of a fully impacted mandibular third molar.

Participants will be randomly assigned to one of four groups:

* Group I (Control): Receive standard care (saline irrigation of the wound).
* Group II (Methylprednisolone): Receive a single 125 mg dose of methylprednisolone intravenously one hour before surgery.
* Group III (Hyaluronic Acid): Receive 2 ml of hyaluronic acid placed directly into the tooth socket after extraction.
* Group IV (Combination): Receive both the pre-operative methylprednisolone injection and the post-extraction hyaluronic acid in the socket.

All participants will receive standard post-operative care, including antibiotics and pain medication, and will be followed up periodically to monitor for complications such as soft tissue issues or infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient medically healthy.
2. Patient between the ages of 18 and 40
3. Patient had impacted mandibular third molar indication for extraction( mesio angler full impaction)
4. Patients who were cooperative, motivated, to attend the follow-up

Exclusion Criteria:

1. Pregnant women, children, elderly (>40 years), physically and mentally challenged, terminally and seriously ill.
2. Patients who had severe pericoronitis, concomitant carious and/or periodontal disease.
3. Patient who had contraindications to the medicines or anesthetics.
4. Uncooperative Patients who won't be able to maintain the follow up visits.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of Post-operative Complications (Pain, Swelling, and Trismus | Baseline (pre-surgery) and at 24 hours, 48 hours, 72 hours, and 7 days post-surgery.

SECONDARY OUTCOMES:
Change in Maximum Interincisal Opening (MIO) | Baseline (pre-surgery) and at 24 hours, 48 hours, 72 hours and 7 days post-surgery.
  Mean Change in Maximum Interincisal Opening (MIO) from Baseline to 7 Days Post-surgery.
  Maximum Interincisal Opening (MIO) is defined as the maximum distance between the incisal edges of the upper and lower central incisors. Measurements will be recorded in millimeters (mm) using a standard surgical ruler. The reported value will be the mean change (decrease or recovery) from the pre-operative baseline measurement at each designated follow-up interval.
  Unit of Measure: Millimeters (mm).
Change in Facial Swelling (Anthropometric Measurement). | Baseline (pre-surgery) and at 24 hours, 48 hours, 72 hours, and 7 days post-surgery
  Mean Change in Facial Swelling (Anthropometric Linear Measurements) Mean Change in Facial Swelling Based on the Sum of Two Linear Distances.
  Facial swelling will be objectively assessed using standardized anthropometric linear measurements (in mm) with a flexible tape or ruler. The total swelling value is calculated as the sum of two distances:
  From the angle of the mouth (Labial Commissure) to the tragus of the ear. From the external canthus of the eye to the angle of the mandible (Gonion). The reported data will be the mean change in the sum of these two distances compared to the pre-operative baseline.
  Unit of Measure: Millimeters (mm).
Incidence of Post-operative Adverse Events. | Baseline (pre-surgery) and at 24 hours, 48 hours, 72 hours, and 7 days post-surgery.
  Number of Participants with Post-operative Adverse Events. This outcome measures the safety and tolerability of the treatment by recording the number of participants who experience any post-operative complications. Adverse events include, but are not limited to: surgical site infection, alveolar osteitis (dry socket), soft tissue dehiscence.
  Unit of Measure: Number of Participants (Count).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Y Al-Eryani, Principal Investigator — Sana'a University
Locations (1):
- Sana'a University, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blondeau F, Daniel NG. Extraction of impacted mandibular third molars: postoperative complications and their risk factors. J Can Dent Assoc. 2007 May;73(4):325. PMID 17484797
- [Background] Altaweel AA, Gaber AE, Alnaffar MZ, Alshomrani EA, Alrehaili RA, Alshaikh RA, Baeshin JN, Al-Akhdar ES. Methylprednisolone and Hyaluronic Acid versus Each Agent Alone to Control Complication of Impacted Wisdom Removal. Evid Based Complement Alternat Med. 2022 Mar 24;2022:1563513. doi: 10.1155/2022/1563513. eCollection 2022. PMID 35368756
- [Background] Alenazi A, Alqhtani NR, Alghannam SS, Alghanim AM, Alasmari M, Almalki S, Eid MK. Effect of Hyaluronic Acid on Socket Healing After Lower Impacted Third Molar Tooth Extraction in 40 Dental Patients. Med Sci Monit. 2024 Sep 16;30:e945386. doi: 10.12659/MSM.945386. PMID 39279207